CLINICAL TRIAL: NCT00995163
Title: Mineral and Bone Disorders Outcomes Study for Japanese Chronic Kidney Disease Stage 5D Patients (MBD-5D)
Brief Title: Mineral and Bone Disorders Outcomes in Stage 5D of Chronic Kidney Disease
Acronym: MBD-5D
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MBD-5D
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: End Stage Renal Disease; Hyperparathyroidism, Secondary
Keywords: outcomes study; hemodialysis; CKD-MBD
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The MBD-5D is a prospective observational study with a case-cohort and a cohort design. Eligible patients are receiving hemodialysis and have secondary hyperparathyroidism. The study's three goals are (1) to record the patients' characteristics, and variation in the patterns of their treatment; (2) to analyze factors associated with variation in those medical practice patterns; and (3) to identify practice patterns and other factors that affect hospitalization, mortality, and other patient-level outcomes.

DETAILED DESCRIPTION:
The MBD-5D is a 3-year prospective observational study with a case-cohort and a cohort design. Eligible patients comprise all patients who are receiving hemodialysis at the participating facilities, and who also have secondary hyperparathyroidism(2HPT). The study has 3 goals: to record the characteristics of those patients and variation in the patterns of their treatment; to analyze factors associated with variation in those medical practice patterns; and to identify the practice patterns and other factors that affect hospitalization, mortality, and other patient-level outcomes. In the case-cohort study, the outcomes are relatively infrequent events (all-cause and cardiovascular mortality). The cohort study includes a randomly selected sample of 40% of all study participants; and the outcomes are hospitalization, parathyroid interventions, bone fracture, MBD management status, etc. Explanatory variables comprise medications and other factors likely to be associated with outcomes of dialysis and of 2HPT, and facility-level practice patterns.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving hemodialysis
* patients whose intact PTH concentration is at least 180 pg/mL (106 pg/mL for whole PTH) OR patients who are receiving intravenous active vitamin D sterols or oral active vitamin D sterols (falecalcitriol)

Exclusion Criteria:

* patients have been undergoing hemodialysis for less than 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who are undergoing hemodialysis and who also have secondary hyperparathyroidism(2HPT)
Sampling Method: Probability Sample
Enrollment: 8020 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 3 years
cardiovascular mortality | 3 years
hospitalization | 3 years

SECONDARY OUTCOMES:
parathyroid interventions | 3 years
bone fracture | 3 years
MBD management status | at 1.5 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tadao Akizawa, MD, PhD, Study Chair — Division of Nephrology, Department of Medicine, Showa University School of Medicine; Masafumi Fukagawa, MD, PhD, Study Director — Division of Nephrology and Metabolism, Tokai University School of Medicine; Shunichi Fukuhara, MD, PhD, Study Director — Department of Epidemiology and Healthcare Research, Graduate School of Medicine, Kyoto University
Locations (1):
- Kobe, Japan

REFERENCES:
- [Derived] Kato C, Fujii N, Miyakoshi C, Asada S, Onishi Y, Fukuma S, Nomura T, Wada M, Fukagawa M, Fukuhara S, Akizawa T. Changes in 3-month mineral and bone disorder patterns were associated with all-cause mortality in prevalent hemodialysis patients with secondary hyperparathyroidism. BMC Nephrol. 2020 Oct 12;21(1):432. doi: 10.1186/s12882-020-02088-x. PMID 33045994
- [Derived] Yamamoto S, Kido R, Onishi Y, Fukuma S, Akizawa T, Fukagawa M, Kazama JJ, Narita I, Fukuhara S. Use of renin-angiotensin system inhibitors is associated with reduction of fracture risk in hemodialysis patients. PLoS One. 2015 Apr 13;10(4):e0122691. doi: 10.1371/journal.pone.0122691. eCollection 2015. PMID 25874620
- [Derived] Fukuhara S, Akizawa T, Fukagawa M, Onishi Y, Yamaguchi T, Hasegawa T, Kurokawa K. Mineral and bone disorders outcomes study for Japanese chronic kidney disease stage 5D patients: rationale and study design. Ther Apher Dial. 2011 Apr;15(2):169-75. doi: 10.1111/j.1744-9987.2010.00906.x. Epub 2011 Mar 2. PMID 21426510